CLINICAL TRIAL: NCT02048319
Title: Assessing Efficacy of Combining Pasireotide With Aspiration Sclerotherapy to Improve Volume Reduction of Dominant Hepatic Cysts: a Randomized, Double-blind, Placebo-controlled Clinical Trial.
Brief Title: Efficacy of Combining Pasireotide With Aspiration Sclerotherapy to Improve Volume Reduction of Hepatic Cysts
Acronym: Sclerocyst
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDTW45115; 2013-003168-29 (EudraCT Number)
Record Dates: First submitted 2014-01-06; First posted 2014-01-29 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Symptomatic Dominant Liver Cyst
Keywords: Liver cyst; Hepatic cyst; Symptomatic; Aspiration sclerotherapy
MeSH Terms: interventions — Injections, Intramuscular; Drainage; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Pasireotide LAR 60 mg (Experimental): The subjects will be randomized (1:1) into two groups. Both groups will undergo aspiration sclerotherapy following the standard procedure. The intervention group will additionally receive two injections of 60 mg pasireotide long-acting release (LAR) intramuscularly: the first injection 14 days before and the second injection 14 days after the intervention.
  Interventions: Drug: Pasireotide LAR 60 mg; Procedure: Aspiration sclerotherapy
- Placebo (Placebo Comparator): Patients in the placebo arm will receive two injections of saline solution corresponding to the scheme of the intervention group.
  Interventions: Procedure: Aspiration sclerotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Pasireotide LAR 60 mg — Pasireotide long acting release, intramuscular injection
  Other Names: Pasireotide long acting release, intramuscular injection
  Arms: Experimental: Pasireotide LAR 60 mg
Procedure: Aspiration sclerotherapy — Percutaneous drainage of the hepatic cyst with subsequent ethanol instillation
  Other Names: Drainage with subsequent ethanol instillation
Drug: Placebo — Saline solution, injected as placebo
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
Liver cysts are fluid filled cavities located in the liver. They are present in 2-11% of the general population, typically not causing any symptoms or complications. However, in a small subset of patients complaints of pain, abdominal fullness and distension, dyspnea and nausea occur.

Currently, aspiration and sclerotherapy is a treatment of choice in symptomatic patients with a large dominant liver cyst. However, studies reported early fluid reaccumulation and relative high recurrence rates of cyst growth after aspiration sclerotherapy ultimately leading to re-interventions. In this respect, somatostatin analogues are promising agents known for its volume reducing effect in patients with polycystic liver disease.

In this study the investigators want to evaluate the effect of combining aspiration sclerotherapy with the multi-receptor binding, long-acting somatostatin analogue Pasireotide.

The investigators hypothesize that administrating pasireotide before and after aspiration sclerotherapy could prevent early fluid reaccumulation and thereby result in a greater reduction of cyst diameter. Moreover, the investigators expect a lower rate of cyst recurrence and subsequently lower need for re-interventions.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are diagnosed with a dominant liver cyst with an indication for aspiration and sclerotherapy are suitable for inclusion in this study.

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age 18 - 70 years
* Indication for aspiration and sclerotherapy
* Providing informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study

ASPIRATION SCLEROTHERAPY RELATED EXCLUSION CRITERIA:

1. Signs of cyst bleeding on ultrasound
2. Signs of cyst infection (elevated CRP and/or leukocytes or temperature exceeding 38 degrees with the exclusion of a different focus)
3. Cyst < 5 cm
4. Coagulopathy (INR > 2 or platelets < 80 x 10^9)
5. Severe co-morbidity contraindicating anesthesia (i.e. ASA 4 classification)

   SOMATOSTATIN TREATMENT RELATED EXCLUSION CRITERIA:
6. Patients with a known hypersensitivity to SST analogues or any component of the pasireotide LAR or SQ formulations
7. Pregnant or nursing women
8. Symptomatic cholecystolithiasis
9. QT interval related exclusion criteria:

   * 9.1 Known (congenital) long QT syndrome or QTcF at screening 470 msec
   * 9.2 Family history of long QT syndrome or idiopathic sudden death
   * 9.3 Uncontrolled or significant cardiac disease including recent myocardial infarction, congestive heart failure, unstable angina or sustained and/or clinically significant cardiac arrhythmias (e.g. bradycardia)
   * 9.4 Risk factors for torsades de pointes: hypokalemia, hypomagnesemia, hypocalcaemia, cardiac failure, clinically significant/symptomatic bradycardia, or high grade AV block
   * 9.5 Patients with concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
   * 9.6 Taking anti-arrhythmic medicinal products or other substances that are known to lead to QT prolongation
10. Uncontrolled diabetes as defined by HbA1C > 64 mmol/ml despite adequate therapy
11. History of pancreatitis
12. Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study treatment

    FURTHERMORE:
13. Use of oral contraception or estrogen supplementation
14. Intervention (i.e. aspiration with or without sclerotherapy or surgical intervention) within six months before baseline
15. Treatment with somatostatin analogues within six months before baseline
16. Any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportional diameter change | 4 weeks
  Proportional change (%) in cyst diameter measured by ultrasound 4 weeks after aspiration sclerotherapy.

SECONDARY OUTCOMES:
Absolute reduction (cm) hepatic cyst | 4 weeks
  Absolute change in cyst diameter measured by ultrasound 4 weeks after aspiration sclerotherapy.
Proportional (%) and absolute cyst reduction (cm) after 12 weeks | 12 weeks
  Proportional (%) and absolute change in cyst diameter measured by ultrasound 12 weeks after aspiration sclerotherapy.
Proportion cyst recurrence | 12 weeks
  > 80% of its original diameter
Symptomatic change and health-related quality of life | 4, 12 weeks and 24 weeks
  Assessment of gastro-intestinal symptoms and health-related quality of life by the GIS- and SF-36 questionnaire respectively
Safety | At week 2, week 4, week 6, week 14 and week 26 after first Pasireotide injection
  Any complications or adverse events reported during procedure or follow-up
Proportional (%) and absolute cyst reduction (cm) after 24 weeks | 24 weeks
  Long term proportional (%) and absolute change in cyst diameter measured by ultrasound 24 weeks after aspiration sclerotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center; Department of Gastroenterology & Hepatology, Nijmegen, Netherlands

REFERENCES:
- [Derived] Wijnands TF, Gevers TJ, Kool LJ, Drenth JP. Aspiration sclerotherapy combined with pasireotide to improve reduction of large symptomatic hepatic cysts (SCLEROCYST): study protocol for a randomized controlled trial. Trials. 2015 Mar 7;16:82. doi: 10.1186/s13063-015-0607-3. PMID 25873132